CLINICAL TRIAL: NCT03584100
Title: The Effect of Pneumatic Tourniquet Use on Upper Extremity Edema Following Axillary Lymph Node Dissection
Brief Title: Effect of Pneumatic Tourniquet on Arm Swelling After Lymph Node Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey Yao, MD, Professor of Orthopaedic Surgery, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-40228; NCI-2018-01125 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRS0075 (Other: OnCore)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy Subject

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Patients with prior axillary lymph node dissection (Experimental): Participants raise their arm for 15 minutes, then wear a tourniquet 8000 inflated for 25 minutes. Hand volume is measured by aqueous volumeter at baseline, after use of the tourniquet and every 5 minutes for 30 minutes, while the arm is placed at a raised on head position, shoulder-level brace position, or at waist in a sling position.
  Interventions: Device: Tourniquet 8000
- Healthy Volunteers (Active Comparator): Participants raise their arm for 15 minutes, then wear a tourniquet 8000 inflated for 25 minutes. Hand volume is measured by aqueous volumeter at baseline, after use of the tourniquet and every 5 minutes for 30 minutes, while the arm is placed at a raised on head position, shoulder-level brace position, or at waist in a sling position.
  Interventions: Device: Tourniquet 8000

INTERVENTIONS:
Device: Tourniquet 8000 — Pneumatic tourniquet with appropriate upper extremity cuff, pressure sensing, and ability to set device at 40 mmHg of pressure
  Other Names: Pneumatic tourniquet

SUMMARY:
The purpose of the proposed study is to evaluate the acute impact of swelling caused by low-pressure tourniquet use in the setting of ipsilateral prior axillary lymph node dissection and the change in swelling reduction following tourniquet use in three limb postures versus healthy volunteers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate reduction in swelling and safety of tourniquet use in patients with prior axillary lymph node dissection

OUTLINE:

Participants raise their arm for 15 minutes, then wear a tourniquet inflated for 25 minutes. Hand volume is measured by aqueous volumeter at baseline, after use of the tourniquet and every 5 minutes for 30 minutes, while the arm is placed at a raised on head position, shoulder-level brace position, or at waist in a sling position.

PROCEDURE:

Participants raise their arm for 15 minutes, then wear a tourniquet 8000 inflated for 25 minutes. Hand volume is measured by aqueous volumeter at baseline, after use of the tourniquet and every 5 minutes for 30 minutes, while the arm is placed at a raised on head position, shoulder-level brace position, or at waist in a sling position.

ELIGIBILITY:
Inclusion Criteria:

* Have previously undergone axillary lymph node dissection
* Or healthy volunteers

Exclusion Criteria:

* Have new-onset lymphedema of the involved limb.
* Infection including cellulitis
* Trauma or planned axillary surgery within 6 months of participation
* Any prior axillary radiation

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Yao, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Tourniquet 8000 Arm: Both arms of participants, ie, auxillary lymph node dissection (ALND) and contralateral (control arm) were evaluated with a low-pressure tourniquet.
Period: Overall Study
Arm/Group | Tourniquet 8000 Arm
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Tourniquet 8000 Arm: Both arms of participants (Auxillary lymph node dissection (ALND) and other contralateral) were used.
Arm/Group | Tourniquet 8000 Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Hand Volume Following Tourniquet Use
Description: Hand volume, as an indicator of limb edema / fluid accumulation, was determined with an aqueous volumeter at rest and for the sling and elevated arm positions 30 minutes after an arm tourniquet was placed. Measurements were taken for the affected arm [ie, after axillary lymph node dissection (ALND)], and the same patient's contralateral arm (control, ie, "other arm").
  The mean values for each arm (affected vs control) of the participant group, before (baseline) and 30 minutes after placement of the pneumatic tourniquet were obtained. The difference represents the effect of tourniquet placement. The outcome is reported as the overall mean difference in hand volume from baseline to 30 minutes after tourniquet placement for the ALND arm (affected arm) and the contralateral arm (control arm), with standard deviation.
  12 patients only.
Time Frame: 30 minutes after tourniquet use
Population: Both arms of all participants were measured and are included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Groups:
- Change in Hand Volume Following Tourniquet Use in Axillary Lymph Node Dissection (ALND) Arm: Mean change in hand volume from baseline to 30 minutes after placement of the pneumatic tourniquet, for axillary lymph node dissection (ALND) arm.
- Change in Hand Volume Following Tourniquet Use in Contralateral Arm: Mean change in hand volume from baseline to 30 minutes after placement of the pneumatic tourniquet, for contralateral control arm.
Arm/Group | Change in Hand Volume Following Tourniquet Use in Axillary Lymph Node Dissection (ALND) Arm | Change in Hand Volume Following Tourniquet Use in Contralateral Arm
Number analyzed (Participants) | 12 | 12
mL
  Mean Difference in Hand Volume, Elevated Position | 15.0 (8.5) | 12.1 (5.4)
  Mean Difference in Hand Volume, Sling Position | 12.5 (8.9) | 7.9 (6.9)

2. Secondary Outcome: Difference in Hand Volume Following Tourniquet Use, Between ALND and Control Limbs
Description: Hand volume, as an indicator of limb edema / fluid accumulation, was determined with an aqueous volumeter 30 minutes after an arm tourniquet was placed and the arm held in sling and elevated arm positions. Measurements were taken for the affected arm [ie, after axillary lymph node dissection (ALND)], and the same patient's contralateral arm (control, ie, "other arm"). Measurements were compared to the participant's contralateral control ("the other arm") in the same positions. The difference represents to effect of ALND on hand volume. The outcome is reported as the absolute change in mean hand volume between the affected and control arms, a number without dispersion.
Time Frame: 30 minutes
Population: Both arms of all participants were measured and are included in the analysis. The reported value is a difference of means, a number without dispersion.
Measure: Number; unit: mL
Units Other Than Participants: hands
Groups:
- Difference in Hand Volume, Axillary Lymph Node Dissection (ALND) vs Contralateral Arms, Elevated: Mean change in hand volume 30 minutes after placement of the pneumatic tourniquet, between axillary lymph node dissection (ALND) arm and contralateral arm, both in the elevated position.
- Difference in Hand Volume, Axillary Lymph Node Dissection (ALND) vs Contralateral Arms, Sling: Mean change in hand volume 30 minutes after placement of the pneumatic tourniquet, between axillary lymph node dissection (ALND) arm and contralateral arm, both in the sling position.
Arm/Group | Difference in Hand Volume, Axillary Lymph Node Dissection (ALND) vs Contralateral Arms, Elevated | Difference in Hand Volume, Axillary Lymph Node Dissection (ALND) vs Contralateral Arms, Sling
Number analyzed (Participants) | 12 | 12
Number analyzed (hands) | 24 | 24
mL | 2.9 | 4.6

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Tourniquet 8000 Arm
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT03584100/Prot_SAP_001.pdf